CLINICAL TRIAL: NCT02655536
Title: A Phase II, Open Label, Multicenter Study of Bevacizumab in Combination With Erlotinib Versus Erlotinib Alone in Patients With EGFR Mutant Non-small Cell Lung Cancer Who Have Brain Metastases
Brief Title: Bevacizumab and Erlotinib in Lung Cancer With Brain Metastases, a Phase II Trial
Acronym: BRILLIANT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201510073MIPB
Record Dates: First submitted 2015-12-24; First posted 2016-01-14 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Brain Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bevacizumab plus erlotinib (Experimental): bevacizumab 15mg/kg every 3 weeks plus erlotinib 150mg per day
  Interventions: Drug: Bevacizumab plus erlotinib
- erlotinib (Active Comparator): erlotinib 150mg per day
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Bevacizumab plus erlotinib — Bevacizumab will be administered at a dose of 15 mg/kg on day 1 of every 3 weeks cycle by IV infusion erlotinib will be give at 150mg orally every day for 21 days of every 3 weeks cycle
  Other Names: avastin plus tarceva
  Arms: bevacizumab plus erlotinib
Drug: Erlotinib — erlotinib will be give at 150mg orally every day for 21 days of every 3 weeks cycle
  Other Names: tarceva
  Arms: erlotinib

SUMMARY:
This is an open-label, randomized, multicenter phase II study conducting in 3 medical centers in Asia. Patients will receive erlotinib in combination with bevacizumab or erlotinib alone. This study will enroll EGFR-mutant NSCLC patients who have asymptomatic brain metastases.

The primary objective is to compare the systemic progression-free survival (PFS) to bevacizumab plus erlotinib versus erlotinib alone in patients with EGFR mutant NSCLC who have asymptomatic brain metastases.

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter phase II study conducting in 3 medical centers in Asia. Patients will receive erlotinib in combination with bevacizumab or erlotinib alone. This study will enroll EGFR-mutant NSCLC patients who have asymptomatic brain metastases.

The primary objective is to compare the systemic progression-free survival (PFS) to bevacizumab plus erlotinib versus erlotinib alone in patients with EGFR mutant NSCLC who have asymptomatic brain metastases.

Patients will be randomized, at a 1:1 ratio, into bevacizumab plus erlotinib group or erlotinib alone group. Compute tomography (CT) or MRI scans will be performed every 6 weeks in the first 12 months since start of investigational drugs, and then performed every 12 weeks. Patients will be followed until documented progression at brain and/or extra-cranial lesions. Patients with intracranial progression only are allowed to continue investigational drugs until a second progression of either intracranial progression or extracranial progression, developed, and the time-to extracranial progression will be determined. In patients with EGFR mutant advanced NSCLC who had brain metastases, it was reported that PFS to erlotinib or gefitinib was 6.6 months(Park et al., 2012). In the current study, it is assumed that the median PFS, both intracranial and extracranial included, is 7 months for erlotinib group alone and is 12.3 months for bevacizumab plus erlotinib group (hazard ratio 0.57) (Seto et al., 2014). 109 patients will be required for analysis in this randomized phase II study. Patients will be stratified according to the EGFR L858R mutation and the EGFR exon 19 deletion mutation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, stage IV (AJCC 7th Edition) non-small cell lung cancer.
* A tumor harboring an EGFR mutation known to be associated with erlotinib sensitivity (exon 19 deletion and L858R)
* Documented brain metastases.
* At least one measure brain lesion and one extracranial lesion
* No emergent operation or radiotherapy is indicated. Patients who have received operation for brain tumor may be enrolled if they have recovered from the operation and there are measurable brain lesions after operation.
* No prior exposure to EGFR inhibitors or anti-angiogenesis therapy including bevacizumab.
* No prior systemic anti-cancer therapy for advanced NSCLC is allowed. -Previous adjuvant or neo-adjuvant treatment for non-metastatic disease is permitted if completed ≥ 6 months before the start of study treatment.
* Written informed consent obtained prior to any screening procedures.

  ≥20 years of age.
* Must have discontinued any previous anti-cancer and investigational therapy for at least 28 days, major operation for at least 28 days with full healing of surgical wounds, or radiotherapy for at least 14 days before study treatment administration, and must have recovered to grade 1 from the adverse effects of such treatment before starting study treatment.
* Life expectancy ≥ 3 months.
* ECOG performance status: 0-1.
* Female patients of child-bearing potential should have a negative pregnancy test.
* Required baseline laboratory status:

Hemoglobin>9g/dL Platelet count≥100x109/L Absolute neutrophil count (ANC)≥1.5x109/L without growth factor support Total bilirubin>1.5x upper limit of normal (ULN) AST/SGOT and/or ALT/SGPT>2.5x ULN Serum creatinine clearance >50 ml/min, by either Cockcroft-Gault formula or by 24-hour urine collection analysis

-Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

* Squamous cell carcinoma
* Unable or unwilling to swallow tablet once daily.
* allergy to erlotinib and/or bevacizumab
* Previous treatment of EGFR inhibitors or anti-angiogenesis therapies.
* History of gross hemoptysis (defined as bright red blood of at least 1/2 teaspoon or 2.5 mL per episode) within 3 months prior to randomization unless definitively treated with surgery or radiation
* Symptomatic CNS metastases which are neurologically unstable or requiring increasing doses of steroids to control the CNS condition.
* CNS bleeding; history or clinical evidence of CNS stroke (hemorrhagic or thrombotic) within the last 6 months
* Chronic daily use of aspirin (>325 mg/day) or other full-dose NSAIDs with anti platelet activity. Treatment with other antiplatelet agents (e.g., dipyridamole, ticlopidine, clopidogrel, and/or cilostazol) is permitted.
* Other baseline laboratory values Uncontrolled hypercalcemia (>11.5 mg/dL) Urinary protein to creatinine ratio >1 (spot urine) Serum creatinine >2.0 ULN
* Radiation therapy within 2 weeks prior to the first dose of study drug. Any persistent side effect of prior radiotherapy must be resolved to grade 1 prior to the first dose of study treatment.
* Any unresolved toxicity from previous anticancer therapy > Grade 1.
* Currently receiving any prohibited medications including vitamins supplements, and herbal supplements.
* Unable to undergo an MRI or contrast CT procedures.
* Active HBV or HCV infection, HBV carrier can be enrolled if HBV DNA titer is low under antiviral treatment.
* Known history of HIV seropositivity. HIV testing is not required as part of this study.
* Undergone a bone marrow or solid organ transplant.
* Another malignancy diagnosed or treated within 5 years, except carcinoma in situ or skin cancer.
* Major surgery within 4 weeks prior to initiating study treatment, excluding the placement of vascular access.
* Cardiac conditions as

  1. Uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy).
  2. myocardial infarction
  3. unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible)
  4. Symptomatic heart failure (NYHA grade II-IV)
  5. Clinically significant peripheral vascular disease, abdominal fistula, gastrointestinal perforation, or intra abdominal abscess
  6. Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy)
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment, pre-existing idiopathic pulmonary fibrosis or any evidence of clinically active interstitial lung disease.
* Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5mIU/mL).
* Women of child-bearing potential, defined as all women physically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 6 months after stopping study drug. Highly effective contraception methods include:

Male or female sterilization or

Combination of any two of the following:

Use oral, injected or implanted hormonal methods of contraception. Placement of an intrauterine device (IUD) or intrauterine system (IUS). Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository).

* Women are considered post-menopausal and not of child baring potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Sexually active males must use a condom during intercourse while taking the drug and for 6 more months after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Any other condition that would, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, unable to swallow medication, social/psychological issues, etc.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | The PFS will be evaluated per RECIST 1.1 criteria every 6 weeks for the first 12 months and then every 12 weeks up to 36 months.
  The PFS will be evaluated from date of randomization until the date of documented progression or the date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
overall survival | The survival will be assessed from date of randomization until the date of death from any cause. The survival will be assessed every 3 weeks up to 36 months.
overall response rate | The response rate will be evaluated per RECIST 1.1 criteria every 6 weeks for the first 12 months and then every 12 weeks up to 36 months.
  The response rate will be evaluated from date of randomization until the date of documented progression or the date of death from any cause, whichever came first.
Time-to-central nervous system (CNS) progression | Time-to-central nervous system(CNS) progression will be evaluated per RECIST 1.1 criteria every 6 weeks for the first 12 months and then every 12 weeks up to 36 months.
  The Time-to- CNS progression will be evaluated from date of randomization until the date of documented CNS progression.
Time to extra-CNS progression | Time to extra-CNS progression will be evaluated per RECIST 1.1 criteria every 6 weeks for the first 12 months and then every 12 weeks up to 36 months.
  The Time-to-extra-CNS progression will be evaluated from date of randomization until the date of documented extra-CNS progression.
The PFS-2 in patients in patients with CNS progression only | The PFS-2 will be evaluated per RECIST 1.1 criteria every 6 weeks for the first 12 months and then every 12 weeks up to 36 months.
  The PFS-2 will be evaluated from date of randomization until the date of second documented progression or the date of death from any cause, whichever came first.
Time to neurological symptom progression | Time to neurological symptom progression will be evaluated every 3 weeks up to 36 months.
  Time to neurological symptom will be assessed from date of randomization until the dated of documented progression of neurological symptom.
Number of participants with treatment-related adverse events as assessed by CTCAE version 4.03 | Treatment-related adverse events will be evaluated from date of randomization until 30 days after discontinuation of the trial. It will be evaluated every 3 weeks up to 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Nationa Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deng Z, Qin Y, Liu Y, Zhang Y, Lu Y. Role of Antiangiogenic Agents Combined With EGFR Tyrosine Kinase Inhibitors in Treatment-naive Lung Cancer: A Meta-Analysis. Clin Lung Cancer. 2021 Jan;22(1):e70-e83. doi: 10.1016/j.cllc.2020.08.005. Epub 2020 Sep 18. PMID 33067126